CLINICAL TRIAL: NCT01355887
Title: A Prospective Randomized Comparative Trial to Compare Pringle Maneuver With Either Infrahepatic Inferior Vena Cava Clamping or Low Central Venous Pressure in Complex Liver Resections
Brief Title: A Trial to Compare Pringle Maneuver With Either Infrahepatic Inferior Vena Cava Clamping or Low Central Venous Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Chen Xiaoping, Hepatic Surgery Center, Tongji Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, China
Other Study IDs: CHENXP003
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2008-01

CONDITIONS: Liver Resection
Keywords: blood loss; hepatectomy; prospective study; PTC
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: No biospecimens
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to better comprehend the benefits and efficacy of portal triad clamping with infrahepatic IVC clamping during complex hepatectomy. A randomized comparative trial was performed to compare PTC(pringle triad clamping) with either infrahepatic IVC clamping or low central venous pressure in complex liver resections.

DETAILED DESCRIPTION:
To better comprehend the benefits and efficacy of portal triad clamping with infrahepatic IVC clamping during complex hepatectomy. A randomized comparative trial was performed to compare PTC with either infrahepatic IVC clamping or low central venous pressure in complex liver resections. 192 consecutive patients were involved in this study and allocated equally to two groups. Preoperative demographic and clinical data, details of surgical procedure, pathologic diagnosis, postoperative course and complications were collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were assessed by preoperative medical imagings to have a high risk of backflow bleeding from the major hepatic veins and the IVC, based on the size and location of the tumor. The tumors were ≥5 cm in diameter and they involved the liver segments 7, 8 and/or the cranial portion of segment 4. These tumors were in close proximity or were compressing, but had not actually invaded, the major hepatic veins or IVC
2. Pugh-Child Grade A
3. Indocyanine green retention rate at 15 minutes (ICGR15) < 10%;
4. acceptable clotting profile (platelet count ≥ 50 ×109/L and prothrombin activity ≥ 60%)
5. no previous liver resection.

Exclusion Criteria:

1. extrahepatic metastases in patients with malignancy;
2. patients who refused to take part in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During the study period, all patients who received liver resections were considered to be included into this study.
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2008-01; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping Chen, Doctor, Study Director — Hepatic Surgery Center, Tongji Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, China
Locations (1):
- Hepatic surgery center, Tong ji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Zhu P, Lau WY, Chen YF, Zhang BX, Huang ZY, Zhang ZW, Zhang W, Dou L, Chen XP. Randomized clinical trial comparing infrahepatic inferior vena cava clamping with low central venous pressure in complex liver resections involving the Pringle manoeuvre. Br J Surg. 2012 Jun;99(6):781-8. doi: 10.1002/bjs.8714. Epub 2012 Mar 2. PMID 22389136